CLINICAL TRIAL: NCT02113657
Title: A Feasibility Study To Determine T-cell Responses To Neoantigens Following Treatment With Ipilimumab In Men With Metastatic Castration-Resistant Prostate Carcinoma
Brief Title: T-Cell Responses to Neoantigens Post Treatment With Ipilimumab in Men With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Stand Up To Cancer (Other); High Impact Clinical Research Support Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0444; NCI-2014-01205 (Registry Identifier: NCI CTRP); SUC2CR-AACR-DT10 (Other: Stand Up to Cancer)
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Castration-resistant prostate cancer; CRPC; Metastatic; Hormone therapy treatment; Androgen deprivation therapy; gonadotropin-releasing hormone; GnRH; Ipilimumab; Yervoy; BMS-734016; MDX010
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab (Experimental): Ipilimumab administered by vein at a dose of 3 mg/kg once every 3 weeks for a total of 4 doses.
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — 3 mg/kg by vein once every 3 weeks for a total of 4 doses.
  Other Names: Yervoy; BMS-734016; MDX010

SUMMARY:
The goal of this clinical research study is to study the impact of ipilimumab on the immune system of patients currently receiving hormone therapy. The safety of these drug combinations will also be studied.

This is an investigational study. Ipilimumab is FDA approved and commercially available for the treatment of melanoma. Its use to treat prostate cancer is investigational.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive ipilimumab by vein over about 90 minutes at Weeks 1, 4, 7, and 10. Your blood pressure will be measured every 30 minutes during the infusion, as well as an hour after you are finished receiving the study drug.

You will continue to receive your current hormone therapy as scheduled.

You will be given standard drugs (such as steroids) to help decrease severe side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

You will have a study visit before each dose of ipilimumab, then every 4 weeks for a total of 3 visits after the last dose of ipilimumab. At each of these visits, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3 tablespoons) and urine will be collected for routine tests. This blood will also be used and to measure your protein, PSA levels.
* Blood (up to 7 tablespoons) and urine will be collected to test for biomarkers. (Weeks 7, 14, and 22 only)
* Blood (about 1½ teaspoons) will be drawn to check your testosterone level. (Week 10 only)
* Blood (up to 10 tablespoons) will be drawn to test your immune system. You will sign a separate consent form for this blood draw.

At Weeks 14 and 22, the following tests and procedures will be performed to check the status of the disease:

* You may have a chest x-ray.
* You will have CT scans or MRIs of the abdomen, pelvis. If the doctor thinks it is needed, you will also have a CT scan of the chest. If a CT scan of the chest is done, a chest x-ray is not required.
* You will have a bone scan.

If the study doctor thinks it is needed, you may have additional bone scans or CT scans or MRIs of the abdomen, pelvis, or chest to check the status of the disease.

Length of Study:

You may receive the study drug for up to 10 weeks. You will remain on study (receiving your standard hormone therapy) for up to a total of 22 weeks. You will be taken off study treatment if you have intolerable side effects, if the disease gets worse, or if you are unable to follow study directions. If you develop certain side effects or have certain side effects for a long period of time, you may be taken off study. The study doctor will let you know if you need to be taken off study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent for this protocol.
2. Agreed to participate in laboratory protocol PA13-0291 for the testing of biomarkers as described in this clinical protocol.
3. Patients included in the study must be >/= 18 years old.
4. Histologically or cytologically confirmed carcinoma of the prostate.
5. Subjects must have metastatic prostate cancer mass tissue collection within 3 months of study entry.
6. Evidence of metastatic disease on previous bone scan, CT scan and/or MRI.
7. Asymptomatic or minimally symptomatic.
8. Tumor progression while on hormone therapy with castrate levels serum testosterone (</= 1.7 nmol/L or 50 ng/dL) defined as biopsy-proven, PSA and/or radiographic criteria according to the Prostate Cancer Working Group 2 (PCWG2).Castrate levels of testosterone must be maintained by surgical or medical means throughout the conduct of the study.
9. ECOG performance status </= 1.
10. Patients must have normal organ and marrow function as defined below: a) WBC >/= 2500/uL.; b) ANC >/= 1000/uL.; c) Platelets >/= 75 x 10^3/uL.; d) Hemoglobin >/= 9 g/dL.; e) Creatinine </= 2.5 x ULN.; f) ALT </= 2.5 x ULN for patients without liver metastases. For patients with liver metastasis ALT </= 5 x ULN is allowed.; g) Bilirubin </= 2.5 x ULN (except for patients with Gilbert's Syndrome, who must have a total bilirubin </= 3mg/dL).
11. Patient agrees to use adequate contraception (barrier method of birth control) prior to study entry, during therapy and up to 3 months after last dose of ipilimumab.

Exclusion Criteria:

1. Treatment with any of the following medications or interventions concomitantly or within 28 days of starting ipilimumab: a.) Systemic corticosteroids. Use of inhaled, intranasal, intra-articular and topical steroids is acceptable, as is a short course (i.e. </= 1 day) of corticosteroids to prevent a reaction to the IV contrast used for CT scans.; b.) External beam radiation therapy or major surgery requiring general anesthetic.; c.) Any systemic therapy for prostate cancer (with the exception of bisphosphonates and RANK-ligand inhibitors for bone metastases which are allowed) including chemotherapy, secondary hormonal therapies (such as megestrol acetate, diethylstilbestrol, ketoconazole, abiraterone, enzalutamide) and non-steroidal anti-androgens (such as bicalutamide, flutamide or nilutamide).; d.) Immune modulators, cytokines or vaccines for the management of cancer or non-cancer-related illnesses.;
2. (Exclusion Criteria #2 Cont.): e.) Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month before any dose of ipilimumab).; f.) Any other investigational product.
3. Use of controlled schedule III controlled substances for cancer-related pain control.
4. Autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.
5. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
6. Patients with known brain metastases.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Known HIV, Hepatitis B, or Hepatitis C.
9. Untreated symptomatic spinal cord compressions.
10. Other malignancies requiring active therapy or known to be associated with altered immune response.
11. Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Impact of Ipilimumab on T Cell Responses to prostate cancer neoantigens in both primary tumor and metastatic sites in men with metastatic CRPC | 10 weeks
  T-cell response to neoantigens defined as: At least a 2-fold increase compared to the response seen against irrelevant control targets, and activating at least 0.1% of cells tested, or at least a 2-fold increase compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Padmanee Sharma, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org